CLINICAL TRIAL: NCT02524886
Title: Deep Brain Stimulation for Patients With Tardive Dyskinesia and or Dystonia. Efficacy and Psychiatric and Cognitive Effects
Brief Title: Deep Brain Stimulation for Patients With Tardive Dyskinesia and or Dystonia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was not possible to recruit and include a sufficient number of patients within the timeframe.
Sponsor: GGZ Centraal (Other)
Collaborators: University Medical Center Groningen (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DBS for TD
Record Dates: First submitted 2015-07-27; First posted 2015-08-17 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Tardive Dyskinesia; Tardive Dystonia
Keywords: Deep Brain Simulation; Psychiatric; Side-effects
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate stimulation (Active Comparator): Patients will be implanted with a Medtronic electorde and Active PC pulse generator for deep brain stimulation at baseline and GPi electric stimulation will start immediately after surgery
  Interventions: Device: GPi DBS with Medtronic electorde and Activa PC pulsegenerator
- Delayed stimulation (Sham Comparator): Patients will be implanted with a Medtronic electorde and Active PC pulse generator for deep brain stimulation at baseline and GPi electric stimulation will start 3 months after surgery
  Interventions: Device: GPi DBS with Medtronic electorde and Activa PC pulsegenerator

INTERVENTIONS:
Device: GPi DBS with Medtronic electorde and Activa PC pulsegenerator — The electric stimulation of 2 leads implanted in the Globus Pallidus internus
  Other Names: DBS; GPi-DBS

SUMMARY:
Rationale: Tardive dyskinesia and dystonia (TDD) are severe side effects of dopamine blocking agents, particularly antipsychotics. Deep brain stimulation (DBS) has shown to be effective in the treatment of TDD in psychiatric patients, but only reported in case reports and small clinical trials and with little attention to possible psychiatric or cognitive complications or positive effect on psychiatric symptoms.

Objective: To assess whether treatment with DBS can reduce or resolve TDD and if DBS can induce beneficial or side-effects in particular psychiatric symptoms.

Study design: A delayed onset double blind randomised controlled trial. Study population: Adult patients with a current or previous psychiatric disorder and antipsychotic induced TDD with a stable psychiatric status during the past 6 months.

Intervention: All patients will be treated with DBS in the posteroventrolateral GPi. The groups will be randomised into immediate stimulation or delayed stimulation after 3 months.

Main study parameters/endpoints: Primary objective, improvement on the movement rating scales BFMDRS. Secondary objectives improvement on the quality of life measured on the SF-36, psychiatric stability as measured on the BPRS and the MADRS and cognitive effects as measured on the MATTIS Dementia Rating Scale, Nederlandse Leestest voor Volwassenen (NLV), 15 word test, Facial Expression of Emotion S+T (FEEST), Groninger Intelligentie Test woordopnoemen (GIT), category and letter fluency test, Trail Making Test part A and B and the Stroop colour and word test

ELIGIBILITY:
Inclusion Criteria:

* Mental competence*
* A current or previous psychiatric illness that has been stable for at least the last six months, meaning no overt psychiatric symptoms or decompensation based on a written report of the clinician that is treating the patient
* Diagnosis of TDD, TDD symptoms developed whilst being treated with dopamine blocking agents or within three months (for oral) or within six months (for depot) after withdrawal (definition international review of neurobiology 98)(6)
* TDD must be present for at least 12 months and impede with physical and or social functioning. In this study that is defined as a score of at least 4 on the disability rating scale of the BFMDRS with at least two items scoring a minimum of two, or one item scoring a 3 or higher.
* BFMDRS >12 at the moment of evaluation
* The patient has proven treatment refractory for all other evidence based TDD treatments:

  * Withdrawal of the dopamine blocking agents or a switch to clozapine and/or quetiapine for at least 3 months
  * Adding tetrabenazine at the maximum tolerated dosage for at least 4 weeks
  * In focal dystonia a trial with Botulinum toxin (at least three sessions)
* The patient fully understands that DBS is not a treatment for the psychiatric disorder and agrees to take his or her psychiatric medication as prescribed by their psychiatrist.

Exclusion Criteria:

* The patient has unrealistic expectations of the possible benefit of DBS or does not fully understand the possible side effects and the likelihood of their occurring.
* The patient is suicidal, a score of ≥4 on item 19 on the BPRS
* Mattis scale for dementia <120
* A score of ≥6 on the Clinical Global Impression scale (CGI) psychiatric severity scale or a BPRS ≥68
* A neurological disease that is the cause of the dyskinesia and/or dystonia
* Use of recreational drugs, such cocaine amphetamine or other drugs that affect TDD, within the last 3 months. Cannabis use within the last 3 months is not considered an exclusion criteria
* Previous DBS or ablative stereotactic brain surgery
* General contraindications for stereotactic surgery and general anaesthesia (e.g. severe hypertension, blood coagulation disorder)
* A seizure disorder that is not sufficiently controlled
* An implanted electronic device
* A language barrier that prevents the patients from understanding the investigators or vice versa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-06-25 (Estimated)

PRIMARY OUTCOMES:
DBS efficacy as measured as the change on the Burke Fahn Marsden Dystonia Rating Scale (BFMDRS) | Entire study, measurement at 0, 3, 6 and 12 months for immediate stimulation group and 0, 3, 6, 9, 15 months for the delayed stimulation group
  The Efficacy of the DBS as measured on the Burke Fahn Marsden Dystonia Rating Scale (BFMDRS)

SECONDARY OUTCOMES:
Psychiatric safety as measured on the Brief Psychiatric Rating Scale (BPRS) and the Montgomery-Åsberg Depression Rating Scale (MADRS) | Entire study, measurement at 0, 1.5, 3, 6 and 12 months for immediate stimulation group and 0, 1.5, 3, 6, 9, 15 months for the delayed stimulation group
  Relaps of a pre-exsisting psychiatric condition or the development of a new psychiatric condition as measured on the Brief Psychiatric Rating Scale (BPRS) and the Montgomery-Åsberg Depression Rating Scale (MADRS)
Cognitive side effects as measured using neuropsychological test battery | Entire study, measurement at 0, 3 and 12 months for immediate stimulation group and 0, 3 and 15 months for the delayed stimulation group
  Cognitive effects of DBS as measured using neuropsychological test battery
Quality of life as measured on the Short Form 36 (SF-36) and the World Health Organiasation Brief Quality of Life Score (WHO-Bref) | Entire study, measurement at 0, 3, 6 and 12 months for immediate stimulation group and 0, 3, 6, 9, 15 months for the delayed stimulation group
  The effect of DBS stimulation on the quality of life as measured on the Short Form 36 (SF-36) and the World Health Organiasation Brief Quality of Life Score (WHO-Bref)

CONTACTS AND LOCATIONS:
Overall Officials: Peter N van Harted, MD, PhD, Principal Investigator — GGZ Centraal
Locations (1):
- Zon en Schild, Amersfoort, Utrecht, Netherlands